CLINICAL TRIAL: NCT03009617
Title: Effectiveness of Web-Based Health Education and Consultation on Health Promotion Behaviors of Adolescents: Randomized Controlled Trial
Brief Title: Effectiveness of Web-Based Health Education and Consultation on Health Promotion Behaviors of Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Gulten Guvenc, Assoc. Prof., Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SBUniversitesi
Record Dates: First submitted 2016-12-24; First posted 2017-01-04 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-12

CONDITIONS: Adolescent Health
Keywords: adolescents; web-based health education; eHealth literacy
MeSH Terms: interventions — Counseling

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): The educational program and counseling Pre-test before intervention Monitoring, education, and consultation through the Web At least two reminders via e-mail or phone message a week The last test after three months The website was closed three months later.
  Interventions: Behavioral: the educational program and counseling
- Control Group (No Intervention): Pre-test No intervention The last test after three months Opening the website to the control group

INTERVENTIONS:
Behavioral: the educational program and counseling — to examine the effectiveness of web-based health education and consultation on health promotion behaviors of adolescents, their e-health literacy, and their information levels.
  Arms: Intervention Group

SUMMARY:
Through the training and consultation program conducted via the web for "health promotion," which is an important part of a school's healthcare, interactive communication methods between school nurses and students were provided. The results of the study showed that web-based education and counseling positively influenced health promotion behaviors of the students, and e-health literacy and their knowledge was increased.

DETAILED DESCRIPTION:
Background: Adolescent is a critical period for many health-risk behaviours, such as alcohol consumption, smoking, having unsafe sex, insufficient exercise, and diet, psychological problems, which can be reduced by targeted web-based health education and consultation interventions. Web-based interventions have advantages in terms of acceptability and accessibility and have shown some study to promote health behaviours and e-Health literacy among adolescents.

Objective: The aims of this study was to examine the effectiveness of web-based health education and consultation on health promotion behaviors (ie, smoking, health responsibility, nutrition, interpersonal relationships, spiritual health, alcohol and substance abuse, positive life outlook, unsafe sex, malnutrition) of adolescents and their e-health literacy.

Methods: This randomized controlled study consisted of 252 adolescents, of whom 120 were in the control group and 132 comprised the intervention group. Sociodemographic characteristics of adolescents, internet usage, Adolescent Lifestyle Questionnaire (ALQ), e-health literacy, and information levels of the adolescents were determined before the intervention. No procedures were applied to the control group. A web-based health education and consultation program designed to promote a healthy lifestyle was applied to the intervention group. The results were re-evaluated three months after the intervention.

The investigators first hypothesis is that adolescents in the intervention (the web-based education and consultation) group would report significantly higher level of well-being ( ie, positive life outlook, stress management, spiritual health and health-related quality of life) and health behaviors (ie, health responsibility, nutrition, exercise ) at 3-month follow-up compared to the control group. Second, it is expected that participants in the intervention group would report a significantly higher level of eHealth literacy and knowledge at 3-month follow-up compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* volunteered to participate in the study,
* students who had not yet started high school education (9th-grade students),
* students who had not participated in the pilot scheme (10th-grade students), students who were not non-final year students at the preparation stage for university (12th-grade students), and 11th-grade students who can use the internet.

Exclusion Criteria:

* students who 9th-grade students,
* students who participated in the pilot scheme (10th-grade students), students who were final year students at the preparation stage for university (12th-grade students), and students who can not use the internet

Ages: 17 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 252 (Actual)
Dates: Start 2014-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
adolescents' health behaviors | 6 months
  Adolescent Lifestyle Questionnaire, Information Assessment Form for the Content of Health Education Program

SECONDARY OUTCOMES:
e-Health Literacy | 6 months
  The Health Literacy Scale

IPD SHARING:
Plan to Share IPD: No